CLINICAL TRIAL: NCT04765787
Title: Clinical Response of Nuberol Forte® for the Pain Management in Musculoskeletal Disorders in Routine Pakistani Practice
Brief Title: Safety & Efficacy of Nuberol Forte® in Pain Management
Acronym: NFORT-EFFECT
Status: Completed | Type: Observational
Sponsor: The Searle Company Limited Pakistan (Industry)
Responsible Party: Sponsor
Other Study IDs: TSCL_NFORT-EFFECT_001
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Musculoskeletal Disorder; Pain Management
Keywords: Musculoskeletal Disorder, Nuberol Forte, Pakistan
MeSH Terms: conditions — Musculoskeletal Diseases; Agnosia | interventions — Orphenadrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Painful musculoskeletal disorders in random order: Nuberol Forte® (Paracetamol 650 mg + Orphenadrine 50 mg) for the symptomatic management of the painful musculoskeletal disorders one tablet three times a day or as per physician discretion or as per severity of pain and treatment duration is 7-10 days
  Interventions: Drug: Combination of Paracetamol 650mg + Orphenadrine 50mg

INTERVENTIONS:
Drug: Combination of Paracetamol 650mg + Orphenadrine 50mg — In routine practice for pain , combination of Paracetamol 650 mg + Orphenadrine 50mg prescribed for 7-10 days with follow up and as per physician discretion
  Other Names: Nuberol Forte

SUMMARY:
The global prevalence of Musculoskeletal disorders (MSD) ranges from 14% to as high as 42%. In addition WHO also estimates that 40% of people over the age of 60 years suffer from MSD and about 80% of the people have had low back pain at some point in their life. In Pakistan, to estimate the prevalence of MSD, there is no data available based on the local population. Locally, studies were conducted on the specific subject pools mainly considering the work related musculoskeletal disorders and backache. However, no real data is available for the symptomatic management of painful musculoskeletal disorders in multiple settings to calculate more generalizable results. So this study is planned and if we found good results then it will help physicians to prescribe the above said medicine to all such cases.

DETAILED DESCRIPTION:
The management of musculoskeletal pain is complex therefore plethora of treatment options are available include non-pharmacological treatments , complementary therapies, and pharmacological interventions. In order to provide optimal care to patients with musculoskeletal pain and ensure the efficient use of healthcare resources, a comprehensive overview of the available evidence for the most effective treatment options for musculoskeletal pain presentations is essential. In this context, an observational study is planned on the efficacy and safety of analgesic combination (i.e Nuberol Forte®). Nuberol Forte® is a combination of muscle relaxant (Orphanedrine) and an analgesic/antipyretic (Paracetamol/Acetaminophen). There are clear indications that the combination of Orphenadrine with Paracetamol may give increased antinociceptive activity and duration of action over and above the use of Orphenadrine or Paracetamol alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a clinical history of painful musculoskeletal disorder from last 1 year
* Patient aged ≥18 and ≤70 years inclusive of either sex
* Patient with ability to understand and sign written informed consent form.

Exclusion Criteria:

* Known hypersensitivity to Nuberol Forte product, the metabolites, or formulation excipients.
* Patients with Glaucoma, prostatic hypertrophy or obstruction at the bladder neck, myasthenia gravis, oesophageal spasm and pyloric or duodenal obstruction.
* Treated with Nuberol Forte to evaluate safety as per approved prescribing information for Nuberol Forte in Pakistan.
* Pregnant (assesed on LMP) or breast feeding women (assessed on interview).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pakistani patients suffering from painful musculoskeletal disorders includes ankle and knee sprains, non-articular low-back pain, painful shoulder lesions (rotator cuff syndrome) and a variety of occupational and sport injuries of the soft tissues in random order. In each case, subjective measures of pain, muscle spasm, stiffness and other symptoms of the musculoskeletal pain will be assessed through Muscle & Joint Measure Scale (MJM). The possible side-effects will be recorded along with other data.The physician will recruit the musculoskeletal patients as per standard practice based on the medical judgment and after review of subject's medical history, results of routine screening, physical and general examination.
Sampling Method: Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of Nuberol Forte from baseline to 2 weeks | 2 weeks
  the pain, muscle spasm and stiffness are assessed by Muscle & Joint Measure scale.
To assess the safety of Nuberol Forte in the cases presenting with Musculoskeletal disorder | 2 weeks
  Safety is monitored from the first dose of the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Asif Mahmood, Dr., Study Director — The Searle Company Limited
Locations (3):
- Pakistan (3):
  - Liaquat National Hospital, Karachi, Sindh
  - Medicare Hospital, Karachi, Sindh
  - Patel Hospital, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duffield SJ, Ellis BM, Goodson N, Walker-Bone K, Conaghan PG, Margham T, Loftis T. The contribution of musculoskeletal disorders in multimorbidity: Implications for practice and policy. Best Pract Res Clin Rheumatol. 2017 Apr;31(2):129-144. doi: 10.1016/j.berh.2017.09.004. Epub 2017 Nov 1. PMID 29224692
- [Background] Palazzo C, Ravaud JF, Papelard A, Ravaud P, Poiraudeau S. The burden of musculoskeletal conditions. PLoS One. 2014 Mar 4;9(3):e90633. doi: 10.1371/journal.pone.0090633. eCollection 2014. PMID 24595187
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Babatunde OO, Jordan JL, Van der Windt DA, Hill JC, Foster NE, Protheroe J. Effective treatment options for musculoskeletal pain in primary care: A systematic overview of current evidence. PLoS One. 2017 Jun 22;12(6):e0178621. doi: 10.1371/journal.pone.0178621. eCollection 2017. PMID 28640822
- [Background] Chou R, Peterson K, Helfand M. Comparative efficacy and safety of skeletal muscle relaxants for spasticity and musculoskeletal conditions: a systematic review. J Pain Symptom Manage. 2004 Aug;28(2):140-75. doi: 10.1016/j.jpainsymman.2004.05.002. PMID 15276195
- [Background] Straube A, Aicher B, Fiebich BL, Haag G. Combined analgesics in (headache) pain therapy: shotgun approach or precise multi-target therapeutics? BMC Neurol. 2011 Mar 31;11:43. doi: 10.1186/1471-2377-11-43. PMID 21453539
- [Background] Hoivik HO, Moe N. Effect of a combination of orphenadrine/paracetamol tablets ('Norgesic') on myalgia: a double-blind comparison with placebo in general practice. Curr Med Res Opin. 1983;8(8):531-5. doi: 10.1185/03007998309109793. PMID 6653131
- [Background] McGuinness BW. A double-blind comparison in general practice of a combination tablet containing orphenadrine citrate and paracetamol ('Norgesic') with paracetamol alone. J Int Med Res. 1983;11(1):42-5. doi: 10.1177/030006058301100109. PMID 6219903
- [Background] Hunskaar S, Donnell D. Clinical and pharmacological review of the efficacy of orphenadrine and its combination with paracetamol in painful conditions. J Int Med Res. 1991 Mar-Apr;19(2):71-87. doi: 10.1177/030006059101900201. PMID 1864455
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Syrjala KL, Yi JC, Artherholt SB, Stover AC, Abrams JR. Measuring musculoskeletal symptoms in cancer survivors who receive hematopoietic cell transplantation. J Cancer Surviv. 2010 Sep;4(3):225-35. doi: 10.1007/s11764-010-0126-x. Epub 2010 May 8. PMID 20454867
- [Background] Hameed MH, Ghafoor R, Khan FR, Badar SB. Prevalence of musculoskeletal disorders among dentists in teaching hospitals in Karachi, Pakistan. J Pak Med Assoc. 2016 Oct;66(Suppl 3)(10):S36-S38. PMID 27895349
- [Background] Rathore FA, Attique R, Asmaa Y. Prevalence and Perceptions of Musculoskeletal Disorders Among Hospital Nurses in Pakistan: A Cross-sectional Survey. Cureus. 2017 Jan 26;9(1):e1001. doi: 10.7759/cureus.1001. PMID 28280654
- See also: National Center for Biotechnology Information. PubChem Database. Acetaminophen, CID=1983, (accessed on May 13, 2019) — https://pubchem.ncbi.nlm.nih.gov/compound/1983
- See also: National Center for Biotechnology; Information. PubChem Database. Orphenadrine, CID=4601 (accessed on May 13, 2019) — https://pubchem.ncbi.nlm.nih.gov/compound/4601